

#### 7.1.2019, version 2

Clinical Trial unique protocol ID 2017/12883-1

# Invitation to participate in the research project "Nutrition and Medication" part I

This is an invitation where we ask if you may be willing to be a participant in a research project concerning nutritional status and medication use among elderly persons receiving home nurse services. The aim of the project is to gain more knowledge about undernutrition in the elderly and the relationship between medication use and nutritional status. This is a part of a Ph.D.-project which will be done in collaboration with the Health Care Service in your municipality.

# What does participation in the project imply for you?

If you accept to participate, a qualified nurse or another health care worker from the Home Nurse Service will visit you at home. She will record data related to eating habits, appetite, possible weight loss, illnesses/diseases, and other factors that may possibly influence your intake of food. You will also be asked about your civil status and if you are living alone or not. Your height and weight will be measured, and a photo of your medicines card will be taken. On that picture, also your name and date of birth will be seen.

# Possible benefits and risks by participation

Participation in this project does not imply any risks for you. When visiting you, we will use approximately 15-20 minutes of your time for collecting the health data mentioned above.

#### Voluntary participation and the possibility to withdraw consent

Participation in the project is voluntary. If you wish to take part, you will need to sign the declaration of consent (on the last page in this letter). At any time and without need for giving reason, you are free to withdraw your consent. This will not have any consequences for future provision of health care. If you decide to withdraw participation in the project, you are also free to demand that your data file in this project can be deleted, unless if your anonymized data have already been analysed or used in scientific publications.

If you at a later point, wish to withdraw your consent or have any questions regarding the project, you can contact Ph.D.-candidate and nursing home physician Mari Fiske, University of Oslo, <u>mari.fiske@medisin.uio.no</u>, telephone 926 67 311.

# What will happen to your personal data concerning health?

Any personal data concerning health that has been recorded about you, will only be used as





#### "Nutrition and Medication I"

#### 7.1.2019, version 2

described in the purpose of the project. You have the right to access information that has been recorded about you and the right to see that any error(s) in the recorded data is/are corrected. You also have the right to know which security measures that have been/will be taken when your personal data concerning health is processed.

All information will be processed and used without your name or personal identification number, or any other information that is directly identifiable to you. Linkage between you and your data concerning health will only be possible via a separate identifier list. Only the researchers, professors Jørund Straand and Anne Moen, and Ph.D.-candidate and nursing home physician Mari Fiske will have access to the list.

# Follow- up project

The research project "Nutrition and Medication" consist of two parts. In the first part we will just describe the nutritional status among the participants living two municipalities. Some of the participants in this first part of the project will later be asked for participation in part II.

#### **Finance**

The project is funded of The Norwegian Research Fund for General Practice and the County Governor in Buskerud, Norway.

# **Approval**

The Regional Committee for Medical and Health Research Ethics has reviewed and approved the Research Project. Reference number 2018/1045.

In accordance with the General Data Protection Regulation the University of Oslo, project manager professor Jørund Straand is independently responsible for ensuring that the processing of your personal health data has a legal foundation. This project has a legal foundation in accordance with the EUs General Data Protection Regulation, article 6 no. 1a, article 9 no. 2a, and with your consent.

You have the right to submit a complaint on the processing of your personal health data to the Norwegian Data Inspectorate.

#### **Contact information**

If you have any questions regarding the research project, you can get in touch with Mari Fiske, University of Oslo, <a href="mailto:mari.fiske@medisin.uio.no">mari.fiske@medisin.uio.no</a>, telephone 926 67 311 Jørund Straand, University of Oslo, <a href="mailto:jorund.staand@medisin.uio.no">jorund.staand@medisin.uio.no</a>, telephone: 928 52 523

Anne Moen, University of Oslo, anne.moen@medisin.uio.no



# "Nutrition and Medication I" 7.1.2019, version 2

| I consent to participating i | n the researc | h project and | d that my pe | rsonal data |
|---|---|---|---|---|
| concerning health can be u | ısed as descri | bed above | | |

| Participant's Signature |
|---|
| Participant's Name (in BLOCK<br>LETTERS) |
| I confirm that I have given information about the research project |
| Signature |
| Role in the research project |
| • |